CLINICAL TRIAL: NCT02082392
Title: Developing New Clinical Management Strategies for Antidepressant Treatments
Brief Title: Developing New Clinical Management Strategies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Bret Rutherford, Clinical Professor, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6652
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Clinical Frequency Management: Placebo (Placebo Comparator): Study visits monthly (Week 0, 4, and 8), with phone visits every other week (Week 2 and 6). Double-blind, placebo-controlled treatment with escitalopram 10mg/day, raised to 20mg/day, if non-responders at week 4.
  Interventions: Drug: Placebo
- Research Frequency Management: Placebo (Placebo Comparator): Weekly study visits, treatment with double-blind, placebo controlled escitalopram 10 mg/day, raised to 20mg/day at week 4 if non-responders.
  Interventions: Drug: Placebo
- Clinical Frequency Management: Escitalopram (Active Comparator): Study visits monthly (Week 0, 4, and 8), with phone visits every other week (Week 2 and 6). Double-blind, placebo-controlled treatment with escitalopram 10mg/day, raised to 20mg/day, if non-responders at week 4.
  Interventions: Drug: Escitalopram
- Research Frequency Management: Escitalopram (Active Comparator): Weekly study visits, treatment with double-blind, placebo controlled escitalopram 10 mg/day, raised to 20mg/day at week 4 if non-responders.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram
  Other Names: Lexapro
  Arms: Clinical Frequency Management: Escitalopram; Research Frequency Management: Escitalopram
Drug: Placebo — A substance or treatment of no intended therapeutic value in a pill form.
  Arms: Clinical Frequency Management: Placebo; Research Frequency Management: Placebo

SUMMARY:
The goal of this study is to develop new methods of administering antidepressant medications that will result in improved drug/placebo separation in randomized controlled trials (RCTs) for Major Depressive Disorder (MDD) and enhanced medication response in open clinical treatment. The highly intensive, weekly visit schedule followed in most antidepressant RCTs radically differs from how antidepressant medications are prescribed in standard clinical practice and is believed to be a major reason why the majority of studies submitted to the Food and Drug Administration (FDA) fail to show a significant difference between medication and placebo. Moreover, a "one size fits all" approach to psychopharmacologic management (i.e., weekly visits for all patients) does not take into account differences between patients that may predispose some individuals to respond positively to frequent follow-up visits, while others may respond negatively or not at all. Clinic visits comprise multiple components that may be therapeutic for depression, including activating patients' behavior, exposing them to medical procedures, permitting social interactions with research staff, and providing supportive meetings with clinicians. Two independent meta-analyses have associated more frequent study visits with increased antidepressant and placebo response as well as decreased separation between medication and placebo. Despite the high costs and potential disadvantages of weekly follow-up visits for patients receiving antidepressant medication, this clinical management strategy has not been studied prospectively to date. It is unknown whether weekly follow-up visits are needed to ensure treatment compliance and patient safety in clinical trials and to what degree contacts with clinicians influence medication and placebo response.

DETAILED DESCRIPTION:
This study utilizes a 2 x 2, double-blind, acute, prospective design randomizing adult outpatients with MDD to "Research Frequency Management" (RFM, weekly study visits) vs. "Community Frequency Management" (CFM, every 4 weeks study visits) and antidepressant medication vs.placebo. Specifying visit frequency as the independent variable in this study has the distinct advantages of being easily operationalized for research purposes avoiding a priori assumptions about which components of study visits influence antidepressant and placebo response (i.e., behavioral activation vs. doctor-patient relationship vs. medical procedures). Close monitoring of all subjects will be assured by telephone evaluations of individuals randomized to CFM at intervals between monthly visits, and additional study contacts will be scheduled as necessary to maintain patient safety (all extra-protocol contacts will be recorded and included as a variable in outcome analyses). Additionally, subjects will be characterized extensively on clinical, demographic, and psychological measures to pilot the study assessment battery and search for predictor variables influencing the effects of contact frequency on medication and placebo response.

ELIGIBILITY:
Inclusion Criteria:

* 1. men and women aged 18-60 years
* 2. diagnosis with Diagnostic and Statistical Manual (DSM) IV Major Depressive Disorder (MDD)
* 3. 24-item Hamilton Rating Scale for Depression (HRSD) score greater than or equal to 18
* 4. capable of providing informed consent and complying with study procedures
* 5. using appropriate contraceptive method if woman of child-bearing age

Exclusion Criteria:

* 1. Current comorbid Axis I DSM IV disorder other than Nicotine Dependence, Adjustment Disorder, or Anxiety Disorder
* 2. diagnosis of substance abuse or dependence (excluding Nicotine Dependence) within the past 12 months
* 3. present or past history of psychosis, psychotic disorder, mania, or bipolar disorder
* 4. baseline HRSD score > 28 or HRSD suicide item > 2
* 5. history of allergic or adverse reaction to escitalopram, or non-response to adequate trial of escitalopram (at least 4 weeks at dose of 20mg) during the current episode
* 6. current treatment with psychotherapy, antidepressants, antipsychotics, or mood stabilizers
* 7. CGI-Severity score of 7 at baseline
* 8. acute, severe, or unstable medical illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment will be coordinated through the Adult and Late Life Depression Research Clinic and will include flyers posted around Columbia University Medical Center (CUMC), information posted on the CUMC internet website, advertisements in local newspapers and on radio stations, and outreach to CUMC clinical staff.
Pre-assignment Details: Interested individuals will contact the ALLDRC coordinator, a telephone screening will take place to identify obviously ineligible subjects. Potentially eligible subjects will be scheduled for an evaluation in the ALLDRC, including a clinical interview by a study clinician (psychiatrist or psychologist) and diagnostic rating by trained rater.
Groups:
- Clinical Frequency Management: Study visits monthly (Week 0, 4, and 8), with phone visits every other week (Week 2 and 6). Double-blind, placebo-controlled treatment with escitalopram 10mg/day, raised to 20mg/day, if non-responders at week 4.
  Escitalopram
- Research Frequency Management: Weekly study visits, treatment with double-blind, placebo controlled escitalopram 10 mg/day, raised to 20mg/day at week 4 if non-responders.
  Escitalopram
Period: Overall Study
Arm/Group | Clinical Frequency Management | Research Frequency Management
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Frequency Management | Research Frequency Management | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11.3) | 48 (0) | 46.67 (8.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression
Description: scale for depressive symptoms administered by trained rater. The HRSD is the standard measure of depression severity for clinical trials of antidepressants and was chosen as the primary outcome measure over other depression rating scales to ensure compatibility of study results with our meta-analyses and ongoing studies of expectancy. Although the HRSD list 21 items, the scoring is based on the first 17 items.
  sum of the scores of the first 17 items (range from 0 to 54): 0-7 = NORMAL 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression >=23 = Very Severe Depression
Time Frame: Baseline week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 2 | 1
units on a scale | 25 (4.24) | 31 (0)

2. Secondary Outcome: Hamilton Anxiety Rating Scale (HARS) 14-item Scale
Description: Scale for anxiety symptoms administered by trained rater. The HARS is a standard measure of anxiety severity in pharmacotherapy studies that has been shown to have acceptable reliability and validity in studies of depressed patients. Each item is scored on a scale of 0 (not present) to 4(severe), with a total score range of 0-56, where <17 indi-cates mild severity, 18-24 mild to moderate severity and25-30 moderate to severe.
Time Frame: Baseline week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 2 | 1
units on a scale | 9.5 (7.78) | 13 (0)

3. Secondary Outcome: CGI Severity and Improvement
Description: scales developed to measure the clinician's view of subjects' global functioning before and after initiating a study medication. The CGI correlates well with other standard outcome measures for depression (e.g., HRSD), is sensitive to change in antidepressant trials, and offers clinically understandable anchor points.
  7-point scale: 0 = Not assessed 4 = Moderately ill
  1 = Normal, not at all ill 5 = Markedly ill 2 = Borderline mentally ill 6 = Severely ill 3 = Mildly ill 7 = Among the most extremely ill patients
Time Frame: Baseline week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 2 | 1
units on a scale | 3 (0) | 4 (0)

4. Secondary Outcome: Treatment Emergent Symptom Scale
Description: rating scale for physical symptoms reported during the study. This is a standard means of recording drug-related adverse effects that will allow us to assess whether contact frequency is associated with differences in side effects among study subjects.
Time Frame: Baseline week
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: California Pharmacotherapy Alliance Scale (CALPAS)-Clinician Version
Description: 24 item Likert scale rating the clinician's assessment of the therapeutic alliance, particularly about medication issues, with the patient. This scale is superior to other therapeutic alliance scales because it is focused on drug treatment and does not contain items specific to psychotherapy. Prior studies using the CALPAS reported an association between therapeutic alliance and outcome, and some studies found alliance mediated the effect of expectancy on depression outcome.
Time Frame: Baseline week
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Blind Assessment-Clinician Version
Description: Rates clinician's guess as to the identity of study medication and the confidence in that guess. This assessment is necessary to document the effectiveness of the study's methods of treatment allocation concealment.
Time Frame: 8 weeks
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Quick Inventory of Depressive Symptoms-Self Report (QIDS-SR) 16 Item Scale
Description: rating scale for depressive symptoms based on DSM criteria. A self-report measure for depressive symptoms is valuable in this study, because it is less susceptible to clinician and rater bias. The QIDS-SR has been increasingly used in antidepressant studies (e.g., STAR*D) due to its equivalent weightings for each symptom item, clearly understandable anchor points, and inclusion of all DSM criteria for depression
Time Frame: 8 Weeks
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Treatment Credibility and Expectancy Scale (CES)
Description: 8 item scale in which subjects rate their impression of the credibility of the treatment and how they estimate their expectation of improvement. The CES is the most widely used measure of expectancy and has demonstrated good psychometric properties in multiple studies. For this study, the primary measure of expectancy will be item 4: "By the end of the treatment period, how much improvement in your depressive symptoms do you think will occur?" (0-100%).
Time Frame: 8 Weeks
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Client Satisfaction Questionnaire 8 (CSQ 8)
Description: self-administered scale with items rating respondents' satisfaction with mental health services they are receiving on a 4 point Likert scale. Use of the CSQ 8 will allow us to determine whether CFM and RFM are associated with differences in participant satisfaction.
Time Frame: 8 Weeks
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Cornell Treatment Preference Index
Description: scale used in mental health studies to document the type and strength of patients' treatment preferences. We will use a modified version in this study asking subjects "Based on your experience and how you feel right now, which of the visit frequencies in this study would be your first choice?" The strength of this preference will be measured on a 5-point Likert scale.
Time Frame: 8 weeks
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Revised Life Orientation Test (LOT-R)
Description: scale developed to assess individual differences in generalized optimism versus pessimism. Degree of optimism on this scale has been correlated with the magnitude of placebo response observed in studies of placebo analgesia, and we will determine whether LOT-R scores moderate effects of therapeutic contact.
Time Frame: 8 weeks
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Schedule for Adaptive and Nonadaptive Personality (SNAP)
Description: this questionnaire is a widely used assessment tool for personality disorders that we will also use to identify predictors of response to varying visit frequency.
Time Frame: 8 weeks
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: California Pharmacotherapy Alliance Scale (CALPAS)-Patient Version
Description: 24 item Likert scale rating the patient's assessment of the therapeutic alliance, particularly about medication issues, with the clinician. This scale is superior to other therapeutic alliance scales because it is focused on drug treatment and does not contain items specific to psychotherapy.
Time Frame: 8 weeks
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Blind Assessment-Patient Version
Description: rates subject's guess as to the identity of study medication and the confidence in that guess. This assessment is necessary to document the effectiveness of the study's methods of treatment allocation concealment.
Time Frame: 8 weeks
Population: Data were not collected
Arm/Group | Clinical Frequency Management | Research Frequency Management
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Clinical Frequency Management | Research Frequency Management
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No